CLINICAL TRIAL: NCT04190524
Title: Sonographic Assessment of Cricoid Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David Kantor, Critical Care Physician, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00033746
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Aspiration; Gastric Contents, Anesthesia; Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Control (Other): Each subject will serve as their own control. The esophagus diameter will be measured on each subject, then cricoid pressure will be applied and the esophagus diameter will again be measured.
  Interventions: Other: Application of cricoid pressure; Other: Application of Left lateral paratracheal pressure

INTERVENTIONS:
Other: Application of cricoid pressure — The study first involves recording a baseline image of the neck anatomy using ultrasound, which is a non-invasive, non-irradiating, non-painful imaging modality. Once the baseline anatomy has been imaged, conventional cricoid pressure will be applied with fingers and/or with the ultrasound probe itself and an image will be recorded. The force applied to the cricoid cartilage will be 30 newtons, as determined by a thin force measurement sensor (Tekscan flexiforce sensor) placed in between the patient's skin and the finger (or ultrasound probe).
Other: Application of Left lateral paratracheal pressure — Next, left lateral paralaryngeal pressure will be applied at the level of the cricoid cartilage with fingers and/or the ultrasound probe itself, and the image will again be recorded. Left lateral paralaryngeal pressure will be 30 newtons, as determined by a thin force measurement sensor placed in between the patient's skin and the finger (or ultrasound probe).

SUMMARY:
Examining the effectiveness of cricoid pressure using ultrasound imaging. Pulmonary aspiration of gastric contents during tracheal intubation, although rare in pediatrics, is a potentially catastrophic complication of anesthesia. Cricoid pressure is applied during rapid sequence induction to occlude the esophagus and prevent aspiration of gastric contents. Accumulating evidence in adults suggests that cricoid pressure often is not effective, either because the esophagus normally lies lateral to the cricoid cartilage, or because downward pressure on the cricoid cartilage laterally displaces (rather than compresses) the esophagus. The investigator proposes to examine the effectiveness of cricoid pressure in children in the peri-operative setting using non-invasive ultrasound imaging. Using this approach, the investigator will investigate the normal anatomical relationship of the esophagus and the cricoid cartilage, as well as how cricoid pressures influences this relationship. Further, the investigator will examine whether alternatives to downward cricoid pressure, such as laterally directed pressure, are more effective at occluding the esophagus.

DETAILED DESCRIPTION:
D. Design and methods

1. Study design This study is interventional study of intubated or sedated children who are in the operating room or admitted to the MSICU (Medical Surgical Intensive Care Unit). The intervention is the application of cricoid pressure and also left lateral paratracheal pressure. The outer diameter and position of the esophagus will be assessed sonographically before and after the intervention is performed. Patients and families will be recruited in person either in the pre-op clinic or in the MSICU.
2. Patient selection and inclusion/exclusion criteria All patients age 0 - 17 years who are on the OR (operating room) schedule and all patients admitted to the MSICU will be screened for this study. Patients in the MSICU will only be included if they are sedated as part of their clinical management.

   Exclusion criteria: 1) history of airway or esophageal malformations (e.g. esophageal atresia or trachea-esophageal fistula) or who have had prior surgical procedures involving the airway or esophagus, 2) known difficult airways, 3) patients with tenuous artificial airways as determined by reviewing the CXR (chest x-ray), 4) patients with abnormal blood flow pattern to the head (e.g. history of right carotid ligation or interruption, known incomplete circle of Willis, known right IJ venous clots or obstruction, 5) patients with left neck CVLs (central venous line), and 6) patients with compromised skin integrity on neck.
3. Description of study treatments or exposures/predictors

   The primary physician/surgeon for each patient will be approached for permission to approach the family for consent.

   For operative patients, the study intervention will be performed following completion of the procedure when the patient is emerging from anesthesia. This is a period of time that often lasts 10s of minutes, has very good pain control, and is asleep. Scanning will be performed when the patient is intubated, to identify landmarks, and then as soon as the patient has been extubated to assess for the effect of cricoid or paratracheal pressure. For patients in the MSICU, the study intervention will be performed on any sedated patient who fulfills inclusion and exclusion criteria.

   The study first involves recording a baseline image of the neck anatomy using ultrasound, which is a non-invasive, non-irradiating, non-painful imaging modality. Once the baseline anatomy has been imaged, conventional cricoid pressure will be applied with fingers and/or with the ultrasound probe itself and an image will be recorded. The force applied to the cricoid cartilage will be 30 newtons, as determined by a thin force measurement sensor (Tekscan flexiforce sensor) placed in between the patient's skin and the finger (or ultrasound probe). Next, left lateral paralaryngeal pressure will be applied at the level of the cricoid cartilage with fingers and/or the ultrasound probe itself, and the image will again be recorded. Left lateral paralaryngeal pressure will be 30 newtons, as determined by a thin force measurement sensor placed in between the patient's skin and the finger (or ultrasound probe).
4. Definition of primary and secondary outcomes/endpoints The primary outcome is a change in esophagus outer diameter following the intervention. The diameter will be assessed in the AP(anteroposterior) plane. In addition, the investigator will also record whether the esophageal mucosa is apposed following the application of pressure. Finally, the investigator will record the position of the esophagus relative to the airway before and after the intervention.
5. Data collection methods, assessments, interventions and schedule Data will be collected at the time of ultrasound and uploaded to a secure REDCap database. Patient specific information will be collected, including age, gender, height, weight, primary diagnosis, and size of endotracheal tube. It is possible that additional covariates may be collected post hoc as necessary to complete analysis.
6. Study timeline Data collection will proceed until the sample size is achieved. Interim data analysis will occur when 50% of the proposed sample size has been achieved.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 0 - 17 years who are on the OR (operating room) schedule and all patients admitted to the MSICU (Medical Surgical Intensive Care Unit) will be screened for this study.
* Patients in the MSICU will only be included if they are sedated as part of their clinical management.

Exclusion Criteria:

* history of airway or esophageal malformations (e.g. esophageal atresia or trachea-esophageal fistula) or who have had prior surgical procedures involving the airway or esophagus
* known difficult airways
* patients with tenuous artificial airways as determined by reviewing the CXR (chest x-ray)
* patients with abnormal blood flow pattern to the head (e.g. history of right carotid ligation or interruption, known incomplete circle of Willis, known right IJ (internal jugular) venous clots or obstruction
* patients with left neck CVLs (Central Venous Line)
* patients with compromised skin integrity on neck

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in esophagus outer diameter following cricoid pressure | 20 minutes
  1. To sonographically assess the diameter of the esophagus before and after application of conventional cricoid pressure
  2. To sonographically asses the diameter of the esophagus before and after application of left lateral paralaryngeal pressure

CONTACTS AND LOCATIONS:
Overall Officials: David Kantor, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No